CLINICAL TRIAL: NCT05122377
Title: QoL and Treatment Compliance for Pre-menopausal Patients With HR+ Breast Cancer Using GnRHa as Ovarian Function Suppression(OFS) Treatment in the Chinese Population: a Real-world Observational Investigation
Brief Title: RWE About QOL and Compliance of Patients With OFS in China
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor Shao, Fudan University
Other Study IDs: 2021-40-2343
Record Dates: First submitted 2021-10-29; First posted 2021-11-16 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Quality of Life; Hormone Receptor-positive Breast Cancer
Keywords: GnRHa; patient-reported QoL; treatment compliance
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance | interventions — Leuprolide; Goserelin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GnRHa 3-month: Patients using GnRHa 3-month depot
  Interventions: Drug: 3M GnRHa
- GnRHa 1-month: Patients using GnRHa 1-month depot
  Interventions: Drug: 1M GnRHa

INTERVENTIONS:
Drug: 3M GnRHa — This was a real world, observational study of adjuvant endocrine therapy with GnRHa for OFS in postoperative, premenopausal women with endocrine responsive breast cancer. Patients will receive treatment per GnRHa commercial label instruction: leuprorelin, goserelin, leuprorelin from local like: acetate microspheres sustained for injection(boennuokang), leuprorelin acetate microspheres for injection(beiyi).
  Other Names: Leuprorelin 11.25mg dosage; TAM; AI
  Groups: GnRHa 3-month
Drug: 1M GnRHa — This was a real world, observational study of adjuvant endocrine therapy with GnRHa for OFS in postoperative, premenopausal women with endocrine responsive breast cancer. Patients will receive treatment per GnRHa commercial label instruction: leuprorelin, goserelin, leuprorelin from local like: acetate microspheres sustained for injection(boennuokang), leuprorelin acetate microspheres for injection(beiyi).
  Other Names: Leuprorelin 3.75mg dosage; Goserelin 3.6mg dosage; TAM; AI
  Groups: GnRHa 1-month

SUMMARY:
The purpose of this study is to assess the patient's feedback from using GnRHa depot formulation in postoperative, premenopausal patients with hormone receptor-positive breast cancer.

DETAILED DESCRIPTION:
This was a real world, observational study of adjuvant therapy with GnRHa for OFS in postoperative, premenopausal women with endocrine responsive breast cancer. This trial is designed to compare patients' QOL and treatment compliance measured by FACT-B and self-administered questionnaires during OFS treatment period. Total score of FACT-B and self-administered questionaries, and change from baseline will be calculated and summarized descriptively. Change from baseline will be compared between GnRHa 3-month and GnRHa 1-month using ANCOVA model with baseline value as a covariate.The number depends on the patients who received questionnaire during 18 months recruitment in planned 10 sites. This analytical plan assumes homogeneity across 10 sites so that strata is not considered.

ELIGIBILITY:
Inclusion Criteria:

Age≥18 years old; Both or either ER+ or PgR+ primary tumor; T1-T3, any N, and M0 according to the TNM classification; Any type of breast surgery (includes breast conserving surgery and breast cancer radical surgery); Any type of preoperative and/or postoperative adjuvant chemotherapy prior to enrollment; History of regular menstruation and not having chemical menopause (FSH≥40 mIU/mL and E2<10 pg/mL) within 12 weeks after completion of the postoperative chemotherapy; Previously using GnRH-a 1M or 3M as OFS treatment for at least one time; Capable of receiving other study drug like Tamoxifen or AI; Eastern Cooperative Oncology Group performance status of Grade 0 or 1.

Exclusion Criteria:

Uncapable of receiving endocrine therapy for any clinical or other reason; Bilateral oophorectomy or ovarian irradiation Inflammatory breast cancer or bilateral breast cancer; Multiple cancers or a history of cancer in other organs; Patients with other non-malignant systemic diseases (cardiovascular, renal, hepatic, lung, etc.) that would prevent prolonged follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Premenopausal patients with histologically confirmed primary breast cancer with OFS treatment
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Quality of life (QOL) | Change will be assessed over two time points (baseline and 3 months)
  QOL of participant will be measured by Functional Assessment of Cancer Therapy -Breast (FACT-B) questionnaires, a 37-item instrument designed to measure five domains of QOL in breast cancer patients. Score range: 0-148. The score includes forward items (the higher score means the better of quality of life) and the reverse items (the higher score means the worse quality of life).
Treatment compliance | Change will be assessed over two time points (baseline and 3 months)
  Treatment compliance will be measured by self-administered questionnaire. Scale score range: 0-40. The score includes forward items (the higher score means the better adherence) and the reverse items (the higher score means the worse adherence).

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China